CLINICAL TRIAL: NCT01637623
Title: Pharmacologic Interventions for Cardiovascular Disease in Obstructive Sleep Apnea
Brief Title: Study of Cardiovascular Disease and Obstructive Sleep Apnea
Acronym: CVD/OSA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2012-0026; U01HL105365 (NIH); A561000 (Other: UW, Madison); PHARM/PHARMACY/PHARMACY (Other: UW, Madison)
Record Dates: First submitted 2012-06-29; First posted 2012-07-11 (Estimated); Results first posted 2020-08-14 (Actual); Last update posted 2020-08-14 (Actual); Status verified 2020-08

CONDITIONS: Severe Obstructive Sleep Apnea (Apnea Hypopnea Index > 30 Events/Hour); Hypertension
Keywords: Hypertension; High Blood Pressure; Sleep Apnea; Obstructive Sleep Apnea; OSA
MeSH Terms: conditions — Sleep Apnea, Obstructive; Hypertension; Sleep Apnea Syndromes | interventions — Losartan; Allopurinol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Losartan (Active Comparator): Losartan 50 mg daily for two weeks, then increased to 100mg daily for 4 weeks if asymptomatic and blood pressure within range.
  Interventions: Drug: Losartan
- Allopurinol (Active Comparator): Allopurinol 300 mg daily for 6 weeks
  Interventions: Drug: Allopurinol
- Placebo (Placebo Comparator): Placebo capsule daily for 6 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Losartan — Losartan 50 mg daily for two weeks, then increased to 100mg daily for 4 weeks if asymptomatic. Remain at 50 mg daily for 4 more weeks or removed from study if symptomatic.
  Arms: Losartan
Drug: Allopurinol — Allopurinol 300 mg daily for 6 weeks
  Arms: Allopurinol
Drug: Placebo — Placebo capsule daily for 6 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if two medicines (allopurinol and losartan) can influence heart and blood vessel health compared to placebo in patients with sleep apnea who are using continuous positive airway pressure (CPAP).

DETAILED DESCRIPTION:
The specific aims of this research project are: 1) Determine if treatment with losartan, an angiotensin type I receptor (AT1R) antagonist, or allopurinol, a XO inhibitor, normalize chemoreflex control of sympathetic outflow and ventilation and improve local vascular regulation and stiffness; and 2) Determine if these interventions reduce the severity of sleep disordered breathing and lower diurnal blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Males and females between ages of 21 and 65 years
* Apnea hypopnea index or respiratory disturbance index greater than or equal to 25 events per hour
* Subjects eligible for CPAP or BiPAP therapy
* Hypertension by clinical history/diagnosis (may be controlled with non- exclusionary medications) or average blood pressure > 140/90 mm Hg (using last two measurements in prior 12 months - or 1 prior blood pressure and 1 blood pressure at screening)

Exclusion Criteria:

* If subject not using CPAP, having AHI > 60 events/hour or oxygen saturation ≤ 65% during sleep
* Presence of clinical CV disease (coronary artery disease, angina, arrhythmias (subjects with sinus arrhythmias will be reviewed by PI for enrollment), stroke, TIA, cor pulmonale, etc.), heart failure, bruits, or diabetes mellitus by clinical diagnosis/history
* Presence of pulmonary disease that results in significant hypoxemia (resting SaO2 < 88%)
* Hypertriglyceridemia (triglycerides >300 mg/dL), diabetes or impaired glucose tolerance (fasting plasma glucose > 125 mg/dL)
* Patients taking angiotensin converting enzyme inhibitors, angiotensin receptor antagonists, potassium-sparing diuretics (without accompanying loop/thiazide diuretic), allopurinol, oxypurinol, febuxostat, amoxicillin, ampicillin, azathioprine or mercaptopurine.
* Patients with chronic kidney disease (Serum creatinine >1.5 mg/dL) or history of significant hyperkalemia (Serum potassium > 5.2 mEq/L) with ARB therapy
* Patients with history of angioedema
* Patients with bilateral,modified radical or radical mastectomies
* Patients who have a Serum potassium > 5.0 mEq/L at the screening visit
* Female patients who are pregnant (determined by urine pregnancy test) or breastfeeding
* Patients with active MRSA or VRE (vancomycin resistant enterococcus) infection
* History of adverse reaction to allopurinol,losartan, or zolpidem**
* Patients who cannot swallow oral capsules
* Patients who are hospitalized or who have been recently hospitalized (last 2 weeks)
* Inability to comply with or complete the protocol or other reasons at the discretion of the investigators

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2012-06; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Dopp, Pharm.D., Principal Investigator — UW Madison School of Pharmacy; Barbara J Morgan, PhD, PT, Principal Investigator — UW Madison School of Medicine
Locations (4):
- United States (4):
  - Aurora Bay Care, Green Bay, Wisconsin
  - Gundersen Lutheran, La Crosse, Wisconsin
  - University of Wisconsin Madison, Madison, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin

REFERENCES:
- [Result] Morgan BJ, Teodorescu M, Pegelow DF, Jackson ER, Schneider DL, Plante DT, Gapinski JP, Hetzel SJ, Dopp JM. Effects of losartan and allopurinol on cardiorespiratory regulation in obstructive sleep apnoea. Exp Physiol. 2018 Jul;103(7):941-955. doi: 10.1113/EP087006. Epub 2018 Jun 8. PMID 29750475

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Losartan | Allopurinol | Placebo
Started | 29 | 30 | 28
Received Intervention | 28 | 30 | 27
Did Not Receive Intervention | 1 | 0 | 1
Analyzed (baseline characteristics data is for the 86 participants analyzed) | 28 | 30 | 28
Completed | 28 | 30 | 25
Not Completed | 1 | 0 | 3
Not completed — Lost to Follow-up | 0 | 0 | 2
Not completed — Physician Decision | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: baseline analysis population includes data for those participants that were analyzed, per the participant flow
Groups:
- Total: Total of all reporting groups
Arm/Group | Losartan | Allopurinol | Placebo | Total
Number analyzed (Participants) | 28 | 30 | 28 | 86
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (12) | 49 (8) | 47 (9) | 49 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 10 | 9 | 34
  Male | 13 | 20 | 19 | 52
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2 | 4
  Not Hispanic or Latino | 27 | 27 | 24 | 78
  Unknown or Not Reported | 0 | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 2 | 3
  White | 27 | 28 | 24 | 79
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 28 | 30 | 28 | 86

OUTCOME MEASURES:

1. Primary Outcome: Change in Muscle Sympathetic Nerve Activity Responses During Hypoxia
Description: The primary outcome variable is the change in the individual slope of the MSNA - SaO2 response curve at 6 weeks and baseline between treatment groups.
Time Frame: baseline and 6 weeks
Population: Data is for fewer subjects than were randomized to treatment because a useable nerve signal was not obtained on all participants.
Measure: Mean (Standard Deviation); unit: bursts/minute*%SaO2
Arm/Group | Losartan | Allopurinol | Placebo
Number analyzed (Participants) | 18 | 23 | 25
bursts/minute*%SaO2
  Baseline | -0.54 (0.29) | -0.84 (0.47) | -0.71 (0.43)
  Following 6 weeks of therapy | -0.69 (.50) | -0.66 (0.38) | -0.61 (0.40)

2. Secondary Outcome: Change in Aortic Pulse Wave Velocity
Description: measurement of vascular stiffness assessed before and after study drug treatment
Time Frame: baseline and 6 weeks
Population: Since this was a secondary outcome measure, not all participants were able to undergo this procedure since scheduling did not always allow with scheduling for primary outcome measure.
Measure: Mean (95% Confidence Interval); unit: m/s
Arm/Group | Losartan | Allopurinol | Placebo
Number analyzed (Participants) | 19 | 20 | 18
m/s | -0.6 [-1.0 to -0.2] | -0.03 [-0.5 to 0.4] | 0.2 [-0.3 to 0.7]

3. Secondary Outcome: Cerebrovascular Conductance
Description: Assessment measures of cerebral blood flow during basal conditions and during graded hypoxia before and after study drug treatment. Cerebrovascular conductance (CVC) was calculated as velocity-time integral/mean arterial pressure.
Time Frame: baseline and 6 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: cm/sec/mmHg
Arm/Group | Losartan | Allopurinol | Placebo
Number analyzed (Participants) | 20 | 20 | 22
cm/sec/mmHg
  baseline | 0.32 (0.13) | 0.27 (0.97) | 0.33 (0.11)
  After six weeks treatment | 0.36 (0.14) | 0.31 (0.12) | 0.34 (0.12)

4. Secondary Outcome: Forearm Vascular Conductance
Description: Assessment measurements of forearm vascular conductance during basal conditions and during graded hypoxia before and after study drug treatment.
Time Frame: baseline and 6 weeks
Population: Participants were not able to conduct all procedures due to scheduling and on occasion, difficulty obtaining a signal. Prioritization of primary outcome measure was the goal.
Measure: Mean (Standard Deviation); unit: ml/min^-1 dL^-1 mmHg^-1
Arm/Group | Losartan | Allopurinol | Placebo
Number analyzed (Participants) | 26 | 30 | 27
ml/min^-1 dL^-1 mmHg^-1
  baseline | 0.41 (0.21) | 0.43 (0.2) | 0.49 (0.31)
  After 6 weeks of treatment | 0.42 (0.17) | 0.55 (0.31) | 0.51 (0.29)

5. Secondary Outcome: Change in Minute Ventilation at Normoxia
Description: assessed before and after study drug treatment
Time Frame: baseline and 6 weeks
Measure: Mean (Standard Deviation); unit: normoxia - L/min
Arm/Group | Losartan | Allopurinol | Placebo
Number analyzed (Participants) | 28 | 30 | 28
normoxia - L/min
  baseline - normoxia in L/min | 8.9 (1.7) | 9.3 (2.1) | 9.3 (2.1)
  six weeks - normoxia in L/min | 8.9 (2.1) | 9.8 (2.6) | 8.8 (1.9)

6. Secondary Outcome: Change in Minute Ventilation During Hypoxia
Description: assessed before and after study drug treatment
Time Frame: baseline and 6 weeks
Measure: Mean (Standard Deviation); unit: hypoxia - L/min*%SaO2
Arm/Group | Losartan | Allopurinol | Placebo
Number analyzed (Participants) | 28 | 30 | 28
hypoxia - L/min*%SaO2
  hypoxia - baseline in L/min*PERCENTSaO2 | -0.41 (0.28) | -0.53 (0.41) | -0.44 (0.29)
  hypoxia - after six weeks treatment in L/min*%SaO2 | -0.37 (0.25) | -0.43 (0.37) | -0.48 (0.32)

7. Secondary Outcome: Aortic Augmentation Index
Description: assessed before and after study drug treatment
Time Frame: baseline and 6 weeks
Population: The number of participants differ between outcome measures due to difficulty in obtaining a viable signal for one outcome vs another and based on scheduling to prioritize the primary outcome measure.
Measure: Mean (95% Confidence Interval); unit: PERCENT of the pulse pressure
Arm/Group | Losartan | Allopurinol | Placebo
Number analyzed (Participants) | 17 | 19 | 14
PERCENT of the pulse pressure
  baseline | 17.3 [12.7 to 22.0] | 18.8 [14.5 to 23.1] | 21.5 [16.8 to 26.3]
  following six weeks of therapy | 16.1 [11.4 to 20.7] | 16.7 [12.5 to 21.0] | 22.5 [17.7 to 27.2]

8. Secondary Outcome: Mean Change in PERCENT Vasodilation
Description: Flow-mediated vasodilation (FMD) (measurement of vascular endothelial function) assessed before and after study drug treatment
Time Frame: baseline and 6 weeks
Population: The number of participants differ between primary and secondary outcome variables due to occasional inability to obtain a viable signal for the variable and due to scheduling difficulties and prioritizing the primary outcome measure.
Measure: Mean (95% Confidence Interval); unit: % change in Max relative FMD
Arm/Group | Losartan | Allopurinol | Placebo
Number analyzed (Participants) | 17 | 19 | 14
% change in Max relative FMD | 1.38 [0.19 to 2.57] | 0.18 [-0.97 to 1.32] | -1.06 [-2.28 to 0.16]

9. Secondary Outcome: Apnea-Hypopnea Index
Description: Severity of sleep apnea assessed before and after study drug treatment
Time Frame: baseline and 6 weeks
Population: as for outcome 8
Measure: Median (Inter-Quartile Range); unit: events/hour
Arm/Group | Losartan | Allopurinol | Placebo
Number analyzed (Participants) | 28 | 28 | 26
events/hour
  baseline | 46 [27 to 58] | 33 [24 to 50] | 35 [18 to 59]
  after six weeks of treatment | 44 [25 to 67] | 45 [22 to 68] | 26 [15 to 62]

10. Secondary Outcome: PERCENT Time Spent Below 88 PERCENT Oxygen Saturation
Description: assessed before and after study drug treatment
Time Frame: baseline and 6 weeks
Population: as for outcome 8
Measure: Median (Inter-Quartile Range); unit: percentage of total sleep time
Arm/Group | Losartan | Allopurinol | Placebo
Number analyzed (Participants) | 28 | 28 | 26
percentage of total sleep time
  baseline | 10 [4 to 25] | 5 [1 to 15] | 5 [1 to 9]
  following six weeks of therapy | 12 [2 to 35] | 8 [2 to 18] | 3 [1 to 8]

11. Secondary Outcome: Change in Mean 24-Hour Blood Pressure (Mean Arterial Pressure)
Description: Change in mean 24 hour blood pressure (mean arterial pressure)
Time Frame: baseline and 6 weeks
Population: as for outcome 8
Measure: Mean (95% Confidence Interval); unit: mm Hg
Arm/Group | Losartan | Allopurinol | Placebo
Number analyzed (Participants) | 23 | 25 | 20
mm Hg | -4.73 [-7.67 to -1.79] | -2.58 [-5.51 to 0.34] | 1.02 [-2.20 to 4.25]

ADVERSE EVENTS:
Time Frame: Up to 6 weeks
Description: Adverse Events Data reported for all participants who started the study, per participant flow.
Arm/Group | Losartan | Allopurinol | Placebo
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/30 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/30 | 0/28
Other Adverse Events (participants affected / at risk) | 0/29 | 0/30 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-25): https://cdn.clinicaltrials.gov/large-docs/23/NCT01637623/Prot_SAP_000.pdf